CLINICAL TRIAL: NCT06226155
Title: TENDAI4PrEP: Adaptation of a Problem-solving Intervention to Address Individual and Provider Level Barriers to PrEP Uptake and Adherence Among Pregnant Women in Zimbabwe
Brief Title: Adaptation of an Intervention Addressing Barriers to PrEP Use Among Pregnant Women in Zimbabwe
Acronym: TENDAI4PrEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Zimbabwe (Other); Boston University (Other)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Director of Behavioral Medicine / Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P003607
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections; Pregnancy Related; Depression, Anxiety
MeSH Terms: conditions — HIV Infections; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENDAI4PrEP (Experimental): TENDAI4PrEP problem-solving intervention will likely entail 4-5 sessions, inclusive of the dyadic session with a partner, with an optional postpartum booster session. The intervention will involve PrEP education and psychoeducation, Nzira Itsva (a culturally adapted Life Steps intervention), and problem-solving therapy.
  Interventions: Behavioral: TENDAI4PrEP
- Enhanced Treatment as Usual (ETAU) (Active Comparator): Participants randomized to ETAU will receive care as usual, which is monthly visits to the ANC, plus a pamphlet of information that describes PrEP efficacy, safety during pregnancy/postpartum, and PrEP availability at the ANC. Antenatal treatment as usual will also be enhanced at the clinic level through the provider-level training, which will be offered to all clinic staff in a nonrandomized design. ETAU participants will also be referred for psychological services at the hospital.
  Interventions: Other: Enhanced treatment as usual

INTERVENTIONS:
Behavioral: TENDAI4PrEP — An adapted problem-solving PrEP use intervention for HIV negative pregnant persons living with psychological distress, their partners, and antenatal care providers.
  Arms: TENDAI4PrEP
Other: Enhanced treatment as usual — Includes monthly visits to the ANC plus a pamphlet of information that describes PrEP efficacy.
  safety during pregnancy/postpartum, and PrEP availability at the ANC.
  Arms: Enhanced Treatment as Usual (ETAU)

SUMMARY:
The purpose of this study is to develop a multi-level PrEP adherence and persistence intervention as an adaptation of the TENDAI ('grateful' in Shona) program, a problem-solving approach to reduce depression and increase HIV treatment adherence among people living with HIV in Zimbabwe. The new intervention, TENDAI4PrEP, will be designed to improve PrEP uptake and persistence among pregnant persons in Zimbabwe. If feasibility, acceptability, and preliminary efficacy are demonstrated, the intervention will be ready for large-scale effectiveness/implementation testing. This program will has the potential to address a critical public health challenge impacting pregnant and postpartum persons in Zimbabwe: the prevention of HIV acquisition and transmission.

DETAILED DESCRIPTION:
Zimbabwe's HIV prevalence rate is among the highest globally, and cisgender women of reproductive age are disproportionately affected. Considering the increased risk of HIV acquisition and transmission during pregnancy, there is an urgent public health need to develop interventions that increase the use of efficacious HIV prevention strategies like PrEP in the antenatal context. Oral pre-exposure prophylaxis (PrEP) is safe during pregnancy, effective in preventing HIV, and available in Zimbabwean antenatal care (ANC) clinics. However, PrEP use remains low among cisgender women of reproductive age. Individual-, interpersonal/community-, and provider-level barriers (e.g., psychological distress, stigma, low partner support, limited PrEP knowledge in providers) compromise use.

A multi-level, problem-solving intervention that addresses barriers to PrEP adherence and persistence during pregnancy and through the postpartum transition among patients, their partners, and antenatal care providers could improve the health of pregnant persons, ultimately decreasing HIV incidence in Zimbabwe.

The aims of this study are as follows:

Aim 1: Explore the impact of intersecting, multi-level barriers on PrEP uptake, adherence, and persistence during pregnancy (n=30), and explore barriers to PrEP provision among antenatal care providers (8-10). In individual interviews with HIV-negative pregnant women with psychological distress (15 PrEP naïve, 15 PrEP experienced), the investigators will probe individual, interpersonal/community, and structural barriers/facilitators. It is anticipated that barriers to uptake, adherence, and persistence may include distress linked to common mental health challenges (e.g., depressed mood, posttraumatic stress) at the individual level; lack of support from partners and providers, stigma, and low PrEP awareness at the interpersonal/community level; and limited access to PrEP care and food insecurity/poverty at the structural level. Among providers, interviews will explore PrEP knowledge, perspectives on HIV prevention during pregnancy, and barriers to prescribing PrEP.

Aim 2: Specify the manual and conduct a small proof-of-concept trial with patients (n=5), their partners (n=5), and providers (n=2). The new manual will teach skills to navigate resources and problem solve the multi-level barriers to PrEP use identified in Aim 1 and will include a group-based training for all providers (education on PrEP during pregnancy, negative PrEP attitudes/stigma, and other barriers to prescribing). Content of the manual will be interactively refined on five participants, their partners, and two providers.

Aim 3a: Evaluate the feasibility and acceptability of the patient-level intervention in a pilot RCT (n=70). PrEP eligible pregnant persons with motivation to initiate PrEP who are experiencing psychological distress will be randomized to either the intervention or to enhanced treatment as usual (mental health referral). Primary outcomes will be feasibility and acceptability; it is hypothesized that the intervention (~4-5 sessions, including one dyadic session with a partner, plus a postpartum booster) will be both feasible and acceptable. Aim 3b: Evaluate the feasibility and acceptability of the provider training (~2 sessions), which will be offered to all providers (n~10) in a nonrandomized design; it is hypothesized that the training will be feasible and acceptable. Aim 3c: Explore perceptions of key implementation outcomes among providers and other administrators (n=15) through individual qualitative exit interviews.

ELIGIBILITY:
Inclusion Criteria:

Across all aims participants must be

1. Pregnant
2. Presenting at the Chitungwiza Central Hospital ANC
3. Aged 15+
4. Willing to provide informed consent or assent
5. Have HIV negative status
6. At risk for HIV acquisition (defined as having a male partner of unknown HIV status, suspicions of partner infidelity, reporting multiple partners, or history of STI and/or recent condomless sexual activity)
7. Score >5 on the Shona Symptom Questionnaire

   For the RCT, eligible participants must also be willing to
8. Initiate PrEP prior to randomization
9. Bring their pregnancy partner (if they are safe doing so).

Exclusion Criteria:

1. Inability to provide informed consent/assent and/or complete procedures in Shona or English
2. Current interfering untreated or unstable mental health condition that precludes functional involvement in the study (e.g., active psychosis, untreated bipolar disorder)

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (patient level) | T3 (5 months post-baseline)
  Assessed by (1) 75% of the participants attended at least half of all treatment sessions (2) 80% of the reviewed treatment sessions addressed all key themes, and (3) 60% of the participants completed the assessments at T2 and T3.
Acceptability (patient level) | T3 (5 months post-baseline)
  Assessed via the brief health care interventions framework questionnaire; on average, at least 75% of the participants rate four or more of the items on the postsession acceptability questionnaires with a 4 or a 5 on the Likert-style scale. Scores vary from 1-5, with a higher score indicating higher acceptability.
Feasibility (provider level) | T3 (5 months post-baseline)
  Feasibility will be demonstrated if (1) at least 70% of the antenatal clinic providers attend the group sessions and (2) a review of the audio recording indicates that all key themes were addressed.
Acceptability (provider level) | T3 (5 months post-baseline)
  Assessed via the brief health care interventions framework questionnaire; the sessions will be deemed acceptable if, on average, at least 75% of the providers rate four or more of the items on the post-session acceptability questionnaires with a 4 or a 5 on the Likert-style scale. Scores vary from 1-5, with a higher score indicating higher acceptability.

SECONDARY OUTCOMES:
Self-reported PrEP adherence (patient level) | T2 (2 months post-baseline)
  Assessed at T2 via an adapted version of the Wilson three-item self-report adherence scale.This is a 0-100 scale with 0 representing the lowest possible adherence and 100 representing the highest adherence.
Psychological distress (patient level) | T2 (2 months post-baseline)
  Measured by the Shona Symptom Questionnaire. Scores from 0-14, with a higher score indicating greater psychological distress.
PrEP persistence (patient level) | T3 (5 months post-baseline)
  Determined via DBS and defined as tenofovir-diphosphate (TVF-DP) concentrations of at least 650 fmol/punch for pregnant women and 1050 fmol/punch for postpartum women, indicative of 7 doses per week over a period of up to eight weeks. This threshold may be adjusted pending new data; pregnancy appears to alter the pharmacokinetics of oral PrEP such that differences in TVF-DP levels may be as great as 30-40% between pregnant and postpartum women.
Change in PrEP knowledge (provider level) | Baseline, T3 (5 months post-baseline)
  Will be assessed in a PrEP-Related Knowledge Scale adapted from the Fenway Institute. Total scores may range from 0-8 with higher scores indicating greater PrEP knowledge. PrEP knowledge will be assessed at baseline and 5 months post-baseline to determine change in knowledge after the intervention.
Change in PrEP stigma (provider level) | Baseline, T3 (5 months post-baseline)
  Will be assessed via an adapted version of the Community PrEP-Related Stigma Scale. Each item is measured on a 1-5 Likert Scale. Scores range from 16-80, with higher scores indicating greater stigma. PrEP stigma will be assessed at baseline and 5 months post-baseline to determine change in stigma after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia M Stanton, PhD, Principal Investigator — Boston University; Walter Mangezi, MD, Principal Investigator — University of Zimbabwe
Locations (1):
- University of Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
In accordance with our DMS plan, de-identified data will be deposited to NIMH Data Archive. This will be available to the research community free of charge. In addition to individual level data, the following materials and tools will be made available to interested individuals following achievement of the main aims of the project: qualitative interview guides, qualitative codebooks, and the TENDAI4PrEP intervention manual.
Supporting Information: Study Protocol, SAP
Time Frame: NDA will make decisions about how long to preserve the data; however, NDA has not deleted any deposited data as to date. Data will be deposited every 6 months.
Access Criteria: Those accessing this dataset must register through NDA and agree to the Terms of Use. Users must agree to not re-disseminate data, use appropriate data citation, and to maintain human subjects' protections. The standard NDA data process allows access for one year and is renewable.